CLINICAL TRIAL: NCT00818064
Title: A Randomised, Double-blind, Placebo-controlled, Single- Dose, Dose-escalation Trial of Anti-IL-20 in Healthy Volunteers and Patients With Rheumatoid Arthritis
Brief Title: Safety and Tolerability of Anti-IL-20 in Healthy Volunteers and Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NN8226-3703; 2008-005529-13 (EudraCT Number); EudraCT No: 2008-005529-13
Record Dates: First submitted 2008-12-30; First posted 2009-01-07 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Inflammation; Rheumatoid Arthritis; Healthy
MeSH Terms: conditions — Inflammation; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- A, HV (Experimental): Dose cohort 1 (3 subjects active, 1 placebo)
  Interventions: Drug: anti-IL-20; Drug: placebo
- B, HV (Experimental): Dose cohort 2 (3 subjects active, 1 placebo)
  Interventions: Drug: anti-IL-20; Drug: placebo
- C, HV (Experimental): Dose cohort 3 (3 subjects active, 1 placebo)
  Interventions: Drug: anti-IL-20; Drug: placebo
- D, HV (Experimental): Dose cohort 4 (3 subjects active, 1 placebo)
  Interventions: Drug: anti-IL-20; Drug: placebo
- E, HV (Experimental): Dose cohort 5 (3 subjects active, 1 placebo)
  Interventions: Drug: anti-IL-20; Drug: placebo
- A, RA (Experimental): Dose cohort 1 (3 subjects active, 1 placebo)
  Interventions: Drug: anti-IL-20; Drug: placebo
- B, RA (Experimental): Dose cohort 2 (3 subjects active, 1 placebo)
  Interventions: Drug: anti-IL-20; Drug: placebo
- C, RA (Experimental): Dose cohort 3 (3 subjects active, 1 placebo)
  Interventions: Drug: anti-IL-20; Drug: placebo

INTERVENTIONS:
Drug: anti-IL-20 — Single s.c. injection (per dose cohort)
  Other Names: NN8226
Drug: placebo — Single s.c. injection (per dose cohort)
  Other Names: NN8226

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to investigate the safety and tolerability of single doses of Anti-IL-20 in healthy volunteers (HV) and patients with rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* For healthy volunteers (HV) the following applies:
* Subjects who are considered to be generally healthy based on assessment of medical history, physical examination and clinical laboratory data at screening, as judged by the Investigator
* Females who are post-menopausal, surgically sterile or of non-child-bearing potential
* For rheumatoid arthritis (RA) patients the following applies:
* A diagnosis of rheumatoid arthritis according to the American College of Rheumatology (ACR1987 classification) of at least three months' duration prior to dosing
* Active RA, characterised by a Disease Activity Score 28 (DAS28) greater than 3.2
* Methotrexate treatment (stable doses of maximally 25.0 mg/week for at least 4 weeks) and concomitant intake of folic acid 1 mg/day or 5 mg/week
* Females who are post-menopausal, surgically sterile or of non-child-bearing potential

Exclusion Criteria:

* For healthy volunteers (HV) the following applies:
* Male subjects who do not accept to use double barrier methods of birth control from first dosing until 3 moths after their last visit
* Body mass index (BMI) below 18.5 or above 35.0 kg/m2
* Clinically significant cardiac or cardiovascular disease
* Abnormal blood pressure and heart rate
* Hepatic insufficiency
* Renal insufficiency
* Positive for humane immunodeficiency virus (HIV)
* Positive for hepatitis B (HBV) or hepatitis C (HCV)
* Lymphoproliferative disease
* History or signs of malignancy (except adequately treated and cured basal or squamous cell carcinoma of the skin or cervical carcinoma in situ occurring more than 12 months prior to dosing)
* History of any autoimmune or current inflammatory conditions including rheumatoid arthritis or any other joint disease
* Active or latent tuberculosis: For tuberculosis unvaccinated subjects detected as a positive Mantoux test. For subjects vaccinated against tuberculosis detected as a positive QuantiFeron-test
* Chronic or ongoing infectious disease requiring systemic anti-infectious treatment within the last 2 weeks prior to administration of trial drug
* Any vaccination within the last month before dosing
* Known active viral, bacterial or fungal infection, including herpes, herpes zoster or cold sores 14 days prior to dosing
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 2 weeks prior to dosing, unless in the opinion of the Investigator the medication will not interfere with the trial procedures or compromise the safety of the subject
* History of or current drug and/or alcohol abuse
* Blood donation within the last 3 months (more than 0.45 L)
* For rheumatoid arthritis (RA) patients the following applies:
* Male subjects who do not accept to use double barrier methods of birth control from first dosing until 3 months after their last visit
* Body mass index (BMI) below 18.5 or above 35.0 kg/m2
* Subjects with chronic inflammatory autoimmune disease other than rheumatoid arthritis (except secondary Sjögren's syndrome)
* History of or current inflammatory joint disease other than rheumatoid arthritis (e.g. gout, psoriatic or reactive arthritis, Lyme's disease, juvenile arthritis)
* Chronic or ongoing infectious disease requiring systemic anti-infectious treatment within the last 2 weeks prior to dosing
* Any vaccination within the last month before dosing
* Known active viral, bacterial or fungal infection, including herpes, herpes zoster or cold sores 14 days prior to administration of trial product
* Lymphoproliferative disease
* History or signs of malignancy (except adequately treated and cured basal or squamous cell carcinoma of the skin or cervical carcinoma in situ occurring more than 12 months prior to dosing)
* Use of selective cyclooxygenase-2 (COX-2) inhibitors within the last 2 weeks prior to randomisation
* Concomitant medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Adverse events, including injection site tolerability | during treatment

SECONDARY OUTCOMES:
Terminal serum half-life (t½) | during treatment
Maximum observed serum concentration (Cmax) | during treatment
Time to reach maximum serum concentration (tmax) | during treatment
Area under the serum concentration-time curve (AUC0-t and AUC) | during treatment
Relevant biomarkers in serum and plasma, as well as synovial fluid (if applicable) | during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Groningen, Netherlands

REFERENCES:
- [Result] Lundblad MS, Overgaard RV, Gothberg M, Fjording MS, Watson E. Clinical pharmacokinetics of the anti-interleukin-20 monoclonal antibody NNC0109-0012 in healthy volunteers and patients with psoriasis or rheumatoid arthritis. Adv Ther. 2015 Mar;32(3):228-38. doi: 10.1007/s12325-015-0191-7. Epub 2015 Mar 7. PMID 25749867
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com